CLINICAL TRIAL: NCT06843031
Title: Evaluation of Perfusion Index in the Identification of Postoperative Shivering After General Anesthesia, a Prospective Study
Brief Title: The Role of Perfusion Index in Defining Postoperative Shivering
Status: Active, not recruiting | Type: Observational
Sponsor: Naime Yalçın (Other)
Responsible Party: Sponsor-Investigator, Naime Yalçın, Specialist Anesthesiology and Reanimation, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: KAEK/2019.05.120
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Shivering; Perfusion Index; General Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Arm inhalation anesthesia: Evaluation of peripheral perfusion index during routine monitoring in patients undergoing surgery by gynecologic oncology under desflurane inhalation anesthesia.
- Arm total intravenous anesthesia: Evaluation of peripheral perfusion index during routine monitoring in patients undergoing surgery by gynecologic oncology under total intravenous anesthesia.

SUMMARY:
The relationship between perfusion index and postanesthetic shivering has been investigated in limited studies. Previous studies have investigated the relationship between postanesthetic shivering after total intravenous anesthesia and perfusion index. The relationship between inhalational anesthesia and postoperative shivering has been investigated, but the role of perfusion index on shivering has also been evaluated in limited studies. Therefore, investigators aimed to investigate whether perianesthetic changes in perfusion index in patients under general anesthesia (inhalation anesthesia and total intravenous anesthesia) correlate with the incidence of postanesthetic shivering and whether they are useful in predicting postanesthetic shivering.

DETAILED DESCRIPTION:
Perioperative hypothermia is generally defined as body temperature below 36.0oC. While classified as mild hypothermia (34.C-36.C), moderate hypothermia (32.C-34.C) and severe hypothermia (<32 °C), the most reliable monitoring sites are: pulmonary artery, distal esophagus, nasopharynx and tympanic membrane. measurements. Within approximately 60-90 minutes after anesthesia induction, body temperature decreases with redistribution of the physiological effect of anesthesia. The incidence of perioperative hypothermia in postoperative patients has been reported to be between 20% and 70%. Even mild hypothermia increases the incidence of wound infection, postoperative ischemic myocardial events, and intraoperative blood loss and prolongs the postoperative recovery period. In the hospital environment, the temperature in the extremities is usually 2 to 4°C cooler than the core temperature, and the skin surface is even colder. Body temperature during surgery is affected by a number of anesthesia-related, surgical, environmental, or patient-related risk factors. Surgical risk factors such as surgical technique, duration of surgery, scope of surgery, procedure and amount of irrigation fluid used are at the forefront. In temperature change, behavioral regulation is the strongest thermoregulatory effector. However, patients under anesthesia cannot activate behavioral responses; thermoregulation is only provided by autonomous mechanisms and external thermal management. Vasoconstriction is the most commonly used autonomous effector mechanism in this process. If vasoconstriction is not sufficient and body temperature drops below a certain threshold, shivering begins. Shivering, an involuntary oscillatory pattern of skeletal muscle activity that increases heat production by up to sixfold, is a compensatory mechanism in this sense. It occurs when the temperature of the preoptic area of the hypothalamus decreases. Shivering increases oxygen consumption, causing lactic acidosis, carbon dioxide production, and catecholamine release, eventually increasing cardiac output, heart rate, and arterial pressure. Studies are continuing on the use of perfusion index (PI) for diagnostic purposes regarding the emergence of tremor. Therefore, PI may help reduce the incidence of postoperative shivering with preoperative precautions and preparations. Perfusion index can be calculated using pulse peripheral perfusion oximetry: expressed as the ratio of the pulsatile signal (arterial blood) to the percentage of the non-pulsatile signal (skin, other tissues and non-pulsatile blood), it is a non-invasive measurement, obtained from the amount of infrared light absorbed. PI simultaneously images peripheral perfusion changes during anesthesia, ıt's a very useful monitorization that can help determine the redistribution of body temperature, the effects of vasodilation and their relationship with anesthesia. Previous prospective studies have shown that patients with low PI values before induction of anesthesia are more likely to develop intraoperative hypothermia. It has been found that under general anesthesia, skin temperature contributes almost 20% to the control of vasoconstriction and postanesthetic shivering threshold. In this study, investigator planned to examine whether perioperatif changes in perfusion index are correlated with the incidence of postoperative shivering and therefore whether perfusion index can predict postoperative shivering for preventive purposes under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 20,
* in the ASA I-II, III
* who were planned to undergo elective surgery

Exclusion Criteria:

* under the age of 20,
* those who did not consent,
* those with mental and/or psychiatric disorders,
* in the ASA IV
* History of allergy to drugs to be used in the study

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was prepared as a prospective study and submitted to the approval of the Health Sciences University Kanuni Sultan Süleyman E.A.H. Ethics Committee Committee. The study includes adult female patients over the age of 20 who underwent elective gynecological oncology operations under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
peripheral perfusion index | From enrollment until the 10th minute after extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)